CLINICAL TRIAL: NCT01981629
Title: The Use of the USCOM Device in Addition to Cardiac Ultrasound in Patients Undergoing Treatment for Undifferentiated Shock
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 12-3496
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Shock
Keywords: Shock; USCOM; Cardiac Ultrasound; Emergency Department
MeSH Terms: conditions — Shock; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Shock: Defined by systolic blood pressure less than 95 mmHg or shock index (heart rate/systolic blood pressure) greater than 0.9
  Interventions: Device: USCOM

INTERVENTIONS:
Device: USCOM — The USCOM device will be used in addition to cardiac ultrasound in patients with shock.

SUMMARY:
Currently, bedside ultrasound (US) is performed routinely in emergency department (ED) patients with undifferentiated shock to help guide resuscitation. Previously, it has never been possible to measure cardiac output on patients in the ED. Our clinical question looks at whether the USCOM device gives clinically relevant information in addition to ED cardiac US in patients with shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients in shock, as defined by systolic blood pressure less than 95 mmHg or shock index (heart rate/systolic blood pressure) greater than 0.9

Exclusion Criteria:

* less than 18 years old
* Pregnant
* Patients in shock due to trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department at an urban county hospital.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | Twice during ED visit, averaging one hour
  Cardiac ultrasound findings will be compared to cardiac index and output from the USCOM device

SECONDARY OUTCOMES:
Patient outcomes | After emergency department visit
  Data will be collected on outcomes of patients including death, length of ICU stay, length of hospital stay, and diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Moore, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States